CLINICAL TRIAL: NCT04217759
Title: Effectiveness of Healthy Lifestyle Intervention on Diabetes Risk Reduction Among Bruneian Young Adults: a Randomised Controlled Trial
Brief Title: Healthy Lifestyle Intervention on Diabetes Risk Reduction Among Bruneian Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Brunei Darussalam (Other)
Responsible Party: Principal Investigator, Alifah Nur'ain Haji Mat Rasil, Principal investigator, Universiti Brunei Darussalam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UBDIHS/13H0621
Record Dates: First submitted 2019-12-27; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Overweight and Obesity; Risk Reduction; Diabetes Mellitus, Type 2
Keywords: social cognitive theory; Type 2 diabetes mellitus; social media; diabetes prevention; lifestyle intervention
MeSH Terms: conditions — Overweight; Obesity; Risk Reduction Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated into two groups: one group with intervention (intervention group) and another group without intervention (control group).
  Intervention group went through a healthy lifestyle intervention using evidence-based SCT strategies emphasising on PA and diet for 12 weeks via face-to-face sessions and social media tools, while the control group only received leaflets on healthy lifestyle with no further guidance.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group went through a healthy lifestyle intervention using evidence-based SCT strategies emphasising on PA and diet for 12 weeks via face-to-face sessions and social media tools (Facebook and WhatsApp)
  Interventions: Behavioral: Healthy lifestyle intervention
- Control group (No Intervention): Control group only received leaflets on healthy lifestyle with no further guidance.

INTERVENTIONS:
Behavioral: Healthy lifestyle intervention — The main goal was to provide knowledge and skills for targeted population in order for them to adapt healthy lifestyle throughout their life. At the end of intervention, participants were expected to be fully equipped with necessary knowledge and fundamental skills in adapting and maintaining healthy lifestyle throughout their life. Gradual improvements were emphasised and at least 5% loss of initial body weight was expected, aiming for at least 0.5% loss in the first month.
  It was divided into three phases (preparation, implementation, maintenance) focusing on PA and diet, in which self-efficacy enhancement and self-regulatory skills were emphasised during the first month of intervention.
  Other Names: Be Healthy Camp
  Arms: Intervention group

SUMMARY:
The general research question posed was 'How effective is a healthy lifestyle intervention using behavioural change strategies in the prevention of Type 2 Diabetes Mellitus (T2DM)?'.

The main aim was to assess the effectiveness of a healthy lifestyle intervention implemented for 12 weeks via face-to-face group sessions and by using social media tools (Facebook and WhatsApp) for young adults at risk of T2DM.

The hypothesis was that this healthy lifestyle intervention may be effective in terms of initiating an increased physical activity (PA) level and a healthy balanced dietary intake resulting in improvements of other T2DM risk factors at 12 weeks.

DETAILED DESCRIPTION:
The specific research question posed was 'Is a healthy lifestyle intervention using Social Cognitive Theory (SCT)-based PA and dietary strategies implemented for 12 weeks through face-to-face group sessions and social media tools effective in the initiation and maintenance of increased PA level and healthy balanced dietary intake, resulting in improvements of T2DM risk score, anthropometrics, metabolic parameters and SCT-related psychosocial factors among Bruneian young adults at risk of T2DM?'.

Study design was two-arm parallel, stratified with simple randomisation, and assessor-blinded randomised controlled trial. Participants were randomly allocated into intervention group and control group. Participants were students and alumni of Universiti Brunei Darussalam and Universiti Teknologi Brunei who were overweight-obese at risk of T2DM with a mean age of 23.1 (2.48) years old. Intervention group went through a healthy lifestyle intervention using evidence-based SCT strategies emphasising on PA and diet for 12 weeks, while the control group only received leaflets on healthy lifestyle with no further guidance. Outcomes measured were changes from baseline at week 0 to post-intervention at week 13 between intervention and control groups. Outcomes were changes in diabetes risk score, anthropometrics, metabolic parameters, PA, dietary intake and SCT-related psychosocial factors, with repeated-measures ANOVA as the main analysis.

ELIGIBILITY:
Inclusion Criteria:

* Bruneian including permanent residents
* BMI from 25.00 to 39.99 kg/m2
* American Diabetes Association (ADA) diabetes risk score of at least 3 and maximum score of 8
* Mentally and physically fit with no chronic conditions
* Without medical conditions that could influence glucose metabolism and insulin resistance
* Answered 'No' to all 6 questions in questionnaire-based pre-exercise risk assessment
* Not actively participating in other healthy lifestyle programmes
* Had access to computer or mobile phone with Internet

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Change in diabetes risk score from week 0 to week 13 | 12 weeks
  Using Finnish Diabetes Risk Score (FINDRISC) questionnaire, with minimum score of 0 and maximum score of 22. Score less than 7 as low risk, 7 to 11 as slightly elevated, 12 to 14 as moderate risk, 15 to 20 as high risk and more than 20 as very high risk.

SECONDARY OUTCOMES:
Change in weight (kg) | 12 weeks
  Using digital weighing scale
Change in weight (%) | 12 weeks
  Using digital weighing scale
Height in cm | At baseline
  Using digital weighing scale
Change in body mass index (BMI) (kg/m2) | 12 weeks
  Calculated with weight and height
Change in waist circumference (WC) (cm) | 12 weeks
  Measured at the midpoint between the lower border of the ribcage and iliac crest with tape measure
Change in hip circumference (HC) (cm) | 12 weeks
  Measured at the largest portion of the buttocks with tape measure
Change in waist-to-hip ratio (WHR) | 12 weeks
  Calculated with WC and HC
Change in fasting blood glucose (FBG) (mmol/l) | 12 weeks
  With finger-pricking and AccuTrend Plus System blood analyses
Change in fasting blood total cholesterol (TC) (mmol/l) | 12 weeks
  With finger-pricking and AccuTrend Plus System blood analyses
Change in fasting blood triglycerides (TG) (mmol/l) | 12 weeks
  With finger-pricking and AccuTrend Plus System blood analyses
Change in systolic blood pressure (SBP) (mmHg) | 12 weeks
  Using OMRON automated blood pressure monitor
Change in diastolic blood pressure (DBP) (mmHg) | 12 weeks
  Using OMRON automated blood pressure monitor
Change in resting heart rate (pulse/min) | 12 weeks
  Using OMRON automated blood pressure monitor
Change in vigorous PA metabolic task (MET) (min/week) | 12 weeks
  Using short-form international PA questionnaire (SF-IPAQ)
Change in moderate PA MET (min/week) | 12 weeks
  Using SF-IPAQ
Change in walking MET (min/week) | 12 weeks
  Using SF-IPAQ
Change in total PA MET (min/week) | 12 weeks
  Using SF-IPAQ
Change in sitting time (hrs/day) | 12 weeks
  Using SF-IPAQ
Change in intake of carbohydrates (servings/day) | 12 weeks
  Using 4-day dietary record
Change in intake of protein (servings/day) | 12 weeks
  Using 4-day dietary record
Change in intake of fruits (servings/day) | 12 weeks
  Using 4-day dietary record
Change in Intake of vegetables (servings/day) | 12 weeks
  Using 4-day dietary record
Change in intake of water in (litres/day) | 12 weeks
  Using 4-day dietary record
Change in motivation score | 12 weeks
  Using University of Rhode Island Change Assessment (URICA) with minimum score of -2 and maximum score of 14. The higher the score, the higher the motivation.
Change in social support (diet) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate better support for eating healthy.
Change in social support (PA) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate better support for exercising
Change in overcoming barriers (PA) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate more capabilities to overcome barriers towards exercising
Change in moral disengagement (diet) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate lack of control in eating
Change in outcome expectations (diet) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate more positive expectations for dieting
Change in outcome expectations (PA) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate more positive expectations for exercising
Change in emotional coping (PA) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate better emotional coping by exercising
Change in self-efficacy (PA) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate better confidence in exercising
Facilitation (PA) score | 12 weeks
  Using social cognitive theory (SCT) constructs scale with minimum score of 1 and maximum score of 4. Higher scores indicate better access to facilities and equipment for exercising

CONTACTS AND LOCATIONS:
Overall Officials: Alifah Nur'ain Haji Mat Rasil, Principal Investigator — University Brunei Darussalam
Locations (1):
- PAPRSB Institute of Health Sciences, Universiti Brunei Darussalam, Brunei, Bandar Seri Begawan, Brunei

IPD SHARING:
Plan to Share IPD: Yes
All collected data was available only within the research team which consisted of supervisors only:
  * Dr Nik Tuah (main supervisor)
  * Dr Mas Rina Wati Hamid (co-supervisor)
  * Assoc Prof Dr Ayub Sadiq (co-supervisor)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Throughout Ph.D. course completion until research publications
Access Criteria: Research team
  * Dr Alifah Nur'ain Haji Mat Rasil (principal investigator)
  * Dr Nik Tuah (main supervisor)
  * Dr Mas Rina Wati Hamid (co-supervisor)
  * Assoc Prof Dr Ayub Sadiq (co-supervisor)